CLINICAL TRIAL: NCT02378233
Title: A Double-blinded Randomised Study of Iodine Supplementation to Lactating Women in an Iodine-sufficient Area in Sweden and Evaluation of Maternal and Neonatal Iodine Levels and Thyroid Function
Brief Title: Iodine Status in Swedish Lactating Women - Effect of Iodine Supplementation in the Thyroid Function of Mother and Infant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Fail to complete the recruitment due to lacking resources
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12012002
Record Dates: First submitted 2015-01-19; First posted 2015-03-04 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Gland; Node; Lactation
Keywords: Iodine; Double-Blind Method; Randomized Controlled Trial
MeSH Terms: conditions — Thyroid Diseases; Breast Feeding | interventions — Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iodine (Experimental): iodine containing multivitamin
  150 ug, 1 tablet daily
  Interventions: Dietary Supplement: iodine
- placebo (Placebo Comparator): placebo, 1 tablet Daily of a non-iodine containing multivitamin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: iodine — The intervention is to give a multivitamin pill including 150 microgram iodine and compare with a multivitamin pill that is not including iodine.
  Arms: iodine
Dietary Supplement: Placebo — Patients are given a non-iodine containing multivitamin tablet
  Arms: placebo

SUMMARY:
The aim of the study is to measure urinary milk iodine concentration (MIC), iodine concentration (UIC), thyroid hormones (TSH, FT4) and thyroperoxidase antibodies (TPOab) in breast-feeding women, and UIC in their nursing infants to determine if the levels are adequate, and to see how they can be influenced by 150 ug daily iodine supplementation in breast-feeding women. The hypothesis is that there is a relative iodine deficiency in this sub-population - lactating women and nursing children-, and that this can be influenced by iodine supplementation. Adequate thyroid hormone and iodine levels are very important for small children, when the plasticity of the brain is greatest.

This is as a prospective, double-blind, placebo-controlled study of 221 mothers and their infants. In parallel, 90 age-matched healthy non-pregnant women are recruited. Mothers are randomized to 150 µg/day iodide supplementation or placebo.

Pregnant women are asked for participation on a visit in pregnancy week 37, at the mother health care (MVC) at Mölnlycke and Skövde. The study will run for approximately 3 months for each individual and begins by sampling A (UIC, TSH, FT4, TPOab) at week 37 of the pregnancy, when mothers also get randomized to 150 µg iodine or placebo. New sampling B (UIC, TSH, FT4, MIC ) is collected when the baby is 3 months old. Thereafter the study is completed. In parallel, 90 healthy non-pregnant, non-lactating women in the same age range are recruited and followed with UIC, TSH, FT4, TPOab for 6 months as a control group. In each case a simple questionnaire is filled and blood is also frozen for future analyses.

DETAILED DESCRIPTION:
Are the mothers to be treated with 150 µg iodide per day during lactation to guarantee normal intake of iodine in breast-milk (MIC) and normal urinary iodine concentration (UIC) in their off-spring?

Purpose and Aim This prospective, placebo-controlled study focus on the question whether lactating mothers shall add 150 µg iodide po to guarantee normal MIC and UIC levels in their children or not, as current iodinating program does not guarantee normal levels in these subgroups

* Primary aim: To compare the MIC and UIC of the children to lactating mothers receiving 150 µg iodide or receiving placebo and compare to WHO recommendations.
* Secondary aim: To study UIC in the mothers during lactation compared to controls.

To study the frequency of thyroid dysfunction in lactating women and whether it differs among patients on 150 µg or placebo.

If the UIC concentration in the children breast fed by mothers receiving placebo is lower than the recommended levels by the WHO and if these levels are normalized with 150 µg iodide to the mother this study will be the supportive study for national authorities in Sweden, Europe and in the world to recommend all lactating mothers to add 150 µg when breast feeding even if the country is judged iodine sufficient.

Survey of the field Iodine deficiency in the nature affects thyroid function The supply of iodine varies in different parts of the world, mainly because of varying levels of iodine in the ground water, different soils and plants, different distribution of sea-food, and dissimilar diary food consumption. In many areas with depleted soils and a long distance to the sea, iodine deficiency (ID) is still a major health problem.

Adequate dietary iodine intake is essential for the production of thyroid hormones. Low iodine intake results in the development of hypothyroidism and goiter. Impaired production of thyroid hormones during pregnancy affects growth and brain development in the progeny. Iodine deficiency in school-age children impairs somatic growth, cognitive performance and motor function.

Iodine insufficiency outside Sweden Iodine deficiency remains a public health problem in 47 countries worldwide. Although most countries worldwide have implemented universal salt iodization , countries like Australia, New Zealand and several European countries have been reporting reoccurring iodine deficiency. Changes in food consumption patterns, legislation not covering processed food and decreased salt consumption impose new challenges in ensuring adequate iodine nutrition in the population.

Iodine sufficiency in Sweden In Sweden, goitre was first described by Carl von Linné in 1747, and in the beginning of the 20th century, goitre was detected in 60% of cases in certain areas (19) and in 18% of the total population . A national survey conducted in 1929 confirmed endemic goitre regions located in the inner or eastern part of the country: these iodine deficient areas were known as the "goitre-belt".

These observations contributed to initiation of the Swedish national iodine fortification program for salt in 1936. Initially, 10 mg of potassium iodide (KI) was added to every kilogram salt. In 1966, this was increased to the current level of 50 mg/kg salt, as goitre was still prevalent in some regions of the country.

The first national evaluation of iodine status in Sweden was performed by our group according to the recommendations of the World Health Organization (WHO). Urinary iodine concentration (UIC) was measured in a representative national sample of children aged 6-12 years: the national median UIC was 125 μg/L, indicating optimal iodine nutrition . However, thyroid volumes were higher in Swedish school children than in the international reference study, which may be an effect from genetic and other environmental factors. Iodine intake is considered optimal in Sweden. These findings underline the importance of regular monitoring of iodine intake, especially concerning the decreased intake of table salt that is likely to follow health campaigns and patients with higher need of iodine may be at risk.

Iodine demands increase during pregnancy and lactating The need of iodine is increased during pregnancy and lactating because of the increased thyroid hormone production and enrichment of iodine in breast-milk. An intake of iodide during pregnancy and breast feeding of 250 µg is recommended compared to 150 µg/day in the normal population. Severe iodine deficiency in the new-borne results in cretinism.

The most critical period except for the prenatal period for the child is the two first years of life when the brain still develops. An enhanced risk period is the first 6 month of life when the child is breast-feeding. During this period the child is depending on the iodine concentration in the milk, which is a direct consequence of the mother iodine nutrition. When the infant starts to eat, iodide is supplied from the food.

Numerous studies have measured both thyroid hormones and MIC in women living in iodine sufficient and insufficient regions, which are summarized in three reviews . Three studies have evaluated iodine nutrition in infants longitudinally , whereas the most recent from New Zealand is the longest; during 6 months maternal and infant iodine status were measured.

In the world and the communities of thyroid disease the question is debated whether or not iodide shall be given to pregnant women. American thyroid Association (ATA) has made a strong recommendation for this in fear the even mild iodine deficiency in small children may affect the brain development negatively. WHO has modified their guidelines of supplementation to whether the nation is regarded iodine sufficient, including sufficient levels in pregnant and lactating women (category 1), where no iodide supplementation is need, or not sufficient. The latter group is divided in two; one group where most patient, but <90%, eat iodinated salt and UIC <100 (category 2) and one group with similarly low UIC but where iodized salt is scarcely used (category 3). An iodine supplement of 150 µg is the recommendation in these countries. However, in 2010 Mulrine et al performed a placebo controlled study the first 6 months postpartum. The mothers were iodine deficient, as New Zealand had not implemented an iodizing program, and were supplemented with 75 or 150 µg/day. Both mother and child had UIC and MIC lower than recommend by the WHO. The authors encourage a study done in the circumstances of iodine sufficiency in the nation.

Data from pregnant and lactating women in Sweden are scares. Two small local studies reports median UIC 145-178 µg/dag and 89 µg/l during pregnancy. More knowledge is needed to judge if Swedish woman shall have and iodine supplementation of 150 µg/day or not during this vulnerable period of life for their children.

Project description Study design This is a prospective, double-blinded placebo-controlled trial of 221 lactating women and their children. Mothers are randomized to 150 µg/day iodine supplementation or placebo for 15 weeks. In parallel 90 healthy female controls are recruited from the same community stratified for age and smoking habits. Patients are included after week 36 in pregnancy by the midwife and urinary iodine concentration (UIC), thyroid hormones levels and thyroperoxidase antibodies (TPO-ab) are assessed and a simple questionnaire is filled in by the pregnant women. Placebo/iodine is started at the same visit (allocation 1:1). At the visit 13 (13±1) weeks postpartum UIC, thyroid hormones levels and thyroperoxidase antibodies (TPO-ab) are assessed in all mothers and a simple questionnaire is filled in. MIC is measured in those who still breast-feed. UIC is measured in babies. At all occasion blood specimens are taken, blood is also frozen for future analyses. Weight and length are registered postnatal in the child.

Study population Patients At the antenatal care unit at Mölnlycke and Skövde Health Care center 221 pregnant women aged 18-40 years will be collected consecutively according to inclusion and exclusion criteria.

Inclusion criteria: Pregnant ≥36 weeks, Singleton pregnancy, Aged 18-40 years, Intend to breast-feed, Agree to take no iodine containing supplements during the study postpartum except for study medication, No current thyroid disease Exclusion criteria: Patient who may not attend to the protocol according to the investiga¬tor's opinion, Plans of another pregnancy within the first 6 months postpartum, Vegans

Controls Controls are collected from a randomized sample attain by the Swedish Tax Agency of premenopausal women from Mölnlycke community. Controls in the same age as the patients are contacted by mail for participation in the study and if smoking habits agree with the corresponding patient they come for an inclusion visit. If interested, the controls are told to stop any other iodine containing supplements 1 week before the first visit. If no answer, a reminding letter is sent after two weeks.

Inclusion criteria: Aged 18-40 years, Agree to take no iodine containing supplements during the study postpartum. No current thyroid disease Exclusion criteria: Controls who may not attend to the protocol according to the investiga¬tor's opinion, Plans pregnancy within the next 6 months, Vegans

Significance If the study proves that supplement of 150 µg iodine to mothers guarantee normal iodine intake in the newborn child contact will be taken with the National Food Agency, the National Board Health and Social welfare and the government to lobbying for a general directives of iodine supplementation to all lactating women.

ELIGIBILITY:
LACTATING WOMAN:

Inclusion Criteria:

* 18-40 years.
* Pregnancy longer than week 36.
* Single Pregnancy.
* Planned breastfeeding.
* No current thyroid disease.
* Agree not to take iodine supplementation except as provided through the study.

Exclusion Criteria:

* Patient who is not expected to adhere to the research protocol. Plans for pregnancy within 6 months after delivery.
* Vegans.

CONTROL WOMAN:

Inclusion Criteria:

* 18-40 years.
* No current thyroid disease.
* Agree not to iodine supplementation during the study.

Exclusion Criteria:

* Patient who is not expected to adhere to the research protocol.
* Plans for pregnancy within 6 months of study entry.
* Vegans.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
milk iodine concentration | 3 months after birth (within 7 days)
urinary iodine concentration in the infant | 3 months after birth (within 7 days)

SECONDARY OUTCOMES:
TSH in the mother | pregnancy week 37
TSH in the mother | 3 months after birth
FT4 in the mother | pregnancy week 37
FT4 in the mother | 3 months after birth
TPOab in the mother | pregnancy week 37
TPOab in the mother | 3 months after birth
urinary iodine concentration in the mother | pregnancy week 37
urinary iodine concentration in the mother | 3 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson Nyström, Ass Prof, Principal Investigator — Center for Endocrinology and Metabolism, SAhlgrenska University Hospital, göteborg, Sweden
Locations (1):
- Health Care center, Mölnlycke, Sweden